CLINICAL TRIAL: NCT04098471
Title: A Randomized Controlled Clinical Trial to Investigate the Effects of Transanal Local Excision Following Radiotherapy for the Treatment of Ultra-low T2N0M0 Rectal Cancer
Brief Title: Simple Transanal Local Excision，Transanal Local Excision Following Radiotherapy Versus Total Mesorectum Excision for the Treatment of the Ultra-low T2N0M0 Rectal Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRSYM201909
Record Dates: First submitted 2019-09-19; First posted 2019-09-23 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Rectal Cancer
Keywords: transanal local excision; T2N0M0
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- single transanal loca excision (Experimental)
  Interventions: Procedure: transanal local excision following radiotherapy
- transanal local excision following radiotherapy (Experimental)
  Interventions: Procedure: transanal local excision following radiotherapy
- total mesorectal excision (Experimental)
  Interventions: Procedure: transanal local excision following radiotherapy

INTERVENTIONS:
Procedure: transanal local excision following radiotherapy — transanal local excision following radiotherapy

SUMMARY:
A randomized controlled clinical trial to compare the short and long term outcomes of simple transanal local excision，transanal local excision following radiotherapy or total mesorectal excision for the treatment of Rectal Cancer

DETAILED DESCRIPTION:
Rectal cancer is one of the most common malignancy worldwide. Currently, surgery is the main treatment for stage I rectal cancer, which has good therapeutic effect. For ultra-low rectal cancer, transanal local excision (TLE) has many advantages over total mesorectal excision (TME), such as less trauma, shorter hospitalization time, lower incidence of complications, protection of sexual function and protection of anal function. At present, transanal local excision has become the recommended operation for the T1N0M0 rectal cancer. However, the risk of lymph node metastasis still occurs in stage I tumors, especially in stage T2 tumors, the lymph node metastasis rate can reach 12% - 29% according to the literature. Salvage TME or chemoradiotherapy should be considered for the presence of positive margin of incision, lymphatic/vascular invasion and poor histological differentiation after transanal local excision. At present, the investigators have consulted a large number of literatures and found that TEM is still lack of sufficient evidence in the treatment of T2N0M0 ultra-low rectal cancer. Some studies believed that local excision combined with adjuvant therapy is safe and reliable, but the evidence is not enough. For ultra-low T2N0M0 rectal cancer, more studies need to be carried out to provide guidance for clinical treatment.

In this study, eligible patients will be randomly allocated to operative operation for rectal cancer either by simple TLE，TLE following radiotherapy or TME. 5-years disease free survival rate, 5-years overall survival rate，local recurrence rate and postoperative quality of life will be recorded. Patients will be followed up every 3 months for 2 year, every 6 months for 3 years postoperatively to study the long term effects.

ELIGIBILITY:
Inclusion Criteria:

1. Preoperative pathology confirmed adenocarcinoma.
2. Preoperative MRI or digital examination of tectum confirmed that the distances from the lower edge of the tumors to the anus were less than 5 cm.
3. The mass is not fixed.
4. Preoperative MRI and rectal EUS indicated that the tumor only invaded muscular layer (T2).
5. No suspicious lymphatic metastasis or distant metastasis was found on preoperative high-resolution CT and MRI.
6. American Society of Anesthesiologists(ASA) grade I-III.
7. Informed consent.
8. No history of familial adenomatous polyposis, ulcerative colitis or Crohn's disease.

Exclusion Criteria:

1. Age<18, or>75.
2. Have other cancer history.
3. The pathology of rectal tumors is non-adenocarcinoma.
4. Multiple primary colorectal tumors.
5. Preoperative CT and MR showed that lymphatic metastasis and distant metastasis could be positive.
6. Pregnant or lactating women.
7. Patients with severe mental disorders.
8. ASA score > 3.
9. Receive other cancer treatments (radiotherapy, chemotherapy).
10. Complication with other intestinal diseases (FAP, HNPCC, active ulcerative colitis or Crohn's disease).
11. The general situation is poor and there are other uncontrollable diseases.
12. Preoperative tumor stage was not T2N0M0.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
5-years disease free survival rate | 5 years

SECONDARY OUTCOMES:
5-years overall survival rate | 5 years
local recurrance rate | 5 years
operative time | 1 day
hospitalization time | 15 days
postoperative quality of life as assessed by EORTC QLQ-C30 questionnaire | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Yueming Sun, PhD, Study Director — The First Affiliated Hospital with Nanjing Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tang J, Zhang Y, Zhang D, Zhang C, Jin K, Ji D, Peng W, Feng Y, Sun Y. Total Mesorectal Excision vs. Transanal Endoscopic Microsurgery Followed by Radiotherapy for T2N0M0 Distal Rectal Cancer: A Multicenter Randomized Trial. Front Surg. 2022 Feb 1;9:812343. doi: 10.3389/fsurg.2022.812343. eCollection 2022. PMID 35178428